CLINICAL TRIAL: NCT02443116
Title: A Phase 2, Randomized, Double-blind, Placebo-controlled Study With Additional Open-label, Single-blind and Placebo-controlled Cohorts to Assess the Safety, Tolerability, and Efficacy of NGM282 in Patients With Nonalcoholic Steatohepatitis
Brief Title: Study of NGM282 in Patients With Nonalcoholic Steatohepatitis (NASH)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NGM Biopharmaceuticals, Inc (Industry)
Collaborators: NGM Biopharmaceuticals Australia Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 15-0105
Record Dates: First submitted 2015-05-11; First posted 2015-05-13 (Estimated); Results first posted 2025-06-26 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Nonalcoholic Steatohepatitis (NASH)
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — aldafermin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (9):
- Cohort 1 - Placebo (Placebo Comparator): Cohort 1 - Placebo
  Interventions: Other: Placebo
- Cohort 1 - NGM282 3mg (Experimental): Cohort 1 - NGM282 3mg
  Interventions: Biological: NGM282
- Cohort 1 - NGM282 6mg (Experimental): Cohort 1 - NGM282 6mg
  Interventions: Biological: NGM282
- Cohort 2 - NGM282 0.3mg (Experimental): Cohort 2 - NGM282 0.3mg
  Interventions: Biological: NGM282
- Cohort 2 - NGM282 1mg (Placebo Comparator): Cohort 2 - NGM282 1mg
  Interventions: Biological: NGM282
- Cohort 2 - NGM282 3mg (Experimental): Cohort 2 - NGM282 3mg
  Interventions: Biological: NGM282
- Cohort 3 - NGM282 1mg (Experimental): Cohort 3 - NGM282 1mg
  Interventions: Biological: NGM282
- Cohort 4 - Placebo (Placebo Comparator): Cohort 4 - Placebo
  Interventions: Other: Placebo
- Cohort 4 - NGM282 1mg (Experimental): Cohort 4 - NGM282 1mg
  Interventions: Biological: NGM282

INTERVENTIONS:
Biological: NGM282
  Arms: Cohort 1 - NGM282 3mg; Cohort 1 - NGM282 6mg; Cohort 2 - NGM282 0.3mg; Cohort 2 - NGM282 1mg; Cohort 2 - NGM282 3mg; Cohort 3 - NGM282 1mg; Cohort 4 - NGM282 1mg
Other: Placebo
  Arms: Cohort 1 - Placebo; Cohort 4 - Placebo

SUMMARY:
The purpose of this study is to determine the safety, tolerability, and efficacy of NGM282 in patients with nonalcoholic steatohepatitis.

ELIGIBILITY:
Inclusion Criteria:

* Males or females, between 18 and 75 years of age, inclusive
* Histologically confirmed NASH diagnosis

Exclusion Criteria:

* Clinically significant acute or chronic liver disease
* Prior liver transplantation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 254 (Actual)
Dates: Start 2015-07-31 (Actual); Primary Completion 2019-12-06 (Actual); Study Completion 2020-01-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: NGM Study Director, Study Director — NGM Biopharmaceuticals, Inc
Locations (22):
- United States (17):
  - NGM Clinical Study Site 922, Chandler, Arizona
  - NGM Clinical Study Site 923, Tucson, Arizona
  - NGM Clinical Study Site 924, Los Angeles, California
  - NGM Clinical Study Site 901, San Diego, California
  - NGM Clinical Study Site 902, Denver, Colorado
  - NGM Clinical Study Site 917, Lakewood Rch, Florida
  - NGM Clinical Study Site 906, Chicago, Illinois
  - NGM Clinical Study Site 918, Kansas City, Missouri
  - NGM Clinical Study Site 903, Durham, North Carolina
  - NGM Clinical Study Site 921, Germantown, Tennessee
  - NGM Clinical Study Site 910, Dallas, Texas
  - NGM Clinical Study Site 920, Rollingwood, Texas
  - NGM Clinical Study Site 909, San Antonio, Texas
  - NGM Clinical Study Site 905, San Antonio, Texas
  - NGM Clinical Study Site 904, Charlottesville, Virginia
  - NGM Clinical Study Site 911, Richmond, Virginia
  - NGM Clinical Study Site 908, Seattle, Washington
- Australia (4):
  - NGM Clinical Study Site 703, Sydney, New South Wales
  - NGM Clinical Study Site 704, Adelaide, South Australia
  - NGM Clinical Study Site 701, Melbourne, Victoria
  - NGM Clinical Study Site 705, Melbourne, Victoria
- NGM Clinical Study Site 916, San Juan, Puerto Rico

REFERENCES:
- [Derived] Alkhouri N, Beyer C, Shumbayawonda E, Andersson A, Yale K, Rolph T, Chung RT, Vuppalanchi R, Cusi K, Loomba R, Pansini M, Dennis A. Decreases in cT1 and liver fat content reflect treatment-induced histological improvements in MASH. J Hepatol. 2025 Mar;82(3):438-445. doi: 10.1016/j.jhep.2024.08.031. Epub 2024 Sep 25. PMID 39326675
- [Derived] Nedrud MA, Chaudhry M, Middleton MS, Moylan CA, Lerebours R, Luo S, Farjat A, Guy C, Loomba R, Abdelmalek MF, Sirlin CB, Bashir MR. MRI Quantification of Placebo Effect in Nonalcoholic Steatohepatitis Clinical Trials. Radiology. 2023 Mar;306(3):e220743. doi: 10.1148/radiol.220743. Epub 2022 Nov 1. PMID 36318027
- [Derived] Sanyal AJ, Ling L, Beuers U, DePaoli AM, Lieu HD, Harrison SA, Hirschfield GM. Potent suppression of hydrophobic bile acids by aldafermin, an FGF19 analogue, across metabolic and cholestatic liver diseases. JHEP Rep. 2021 Feb 19;3(3):100255. doi: 10.1016/j.jhepr.2021.100255. eCollection 2021 Jun. PMID 33898959
- [Derived] Loomba R, Ling L, Dinh DM, DePaoli AM, Lieu HD, Harrison SA, Sanyal AJ. The Commensal Microbe Veillonella as a Marker for Response to an FGF19 Analog in NASH. Hepatology. 2021 Jan;73(1):126-143. doi: 10.1002/hep.31523. Epub 2020 Dec 11. PMID 32794259
- [Derived] Harrison SA, Neff G, Guy CD, Bashir MR, Paredes AH, Frias JP, Younes Z, Trotter JF, Gunn NT, Moussa SE, Kohli A, Nelson K, Gottwald M, Chang WCG, Yan AZ, DePaoli AM, Ling L, Lieu HD. Efficacy and Safety of Aldafermin, an Engineered FGF19 Analog, in a Randomized, Double-Blind, Placebo-Controlled Trial of Patients With Nonalcoholic Steatohepatitis. Gastroenterology. 2021 Jan;160(1):219-231.e1. doi: 10.1053/j.gastro.2020.08.004. Epub 2020 Aug 8. PMID 32781086
- [Derived] Harrison SA, Rinella ME, Abdelmalek MF, Trotter JF, Paredes AH, Arnold HL, Kugelmas M, Bashir MR, Jaros MJ, Ling L, Rossi SJ, DePaoli AM, Loomba R. NGM282 for treatment of non-alcoholic steatohepatitis: a multicentre, randomised, double-blind, placebo-controlled, phase 2 trial. Lancet. 2018 Mar 24;391(10126):1174-1185. doi: 10.1016/S0140-6736(18)30474-4. Epub 2018 Mar 5. PMID 29519502

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 254 participants who met all inclusion criteria and no exclusion criteria were enrolled in this study. This was a 3-part study where Parts 1 and 3 were randomized, placebo controlled studies and Part 2 was an open-label study.
Groups:
- Part 1: Aldafermin 3.0 mg: Participants who were randomized to receive a single subcutaneous injection of aldafermin 3.0 mg. The first dose (Day 1) and doses at Weeks 1, 2, 4, 8, and 12 were self-administered in the clinic, with all other doses through Week 12 self-administered at home.
- Part 1: Aldafermin 6.0 mg: Participants who were randomized to receive a single subcutaneous injection of aldafermin 6.0 mg. The first dose (Day 1) and doses at Weeks 1, 2, 4, 8, and 12 were self-administered in the clinic, with all other doses through Week 12 self-administered at home.
- Part 1: Placebo; Part 3: Placebo: Participants who were randomized to receive a single subcutaneous injection of placebo. The first dose (Day 1) and doses at Weeks 1, 2, 4, 8, and 12 were self-administered in the clinic, with all other doses through Week 12 self-administered at home.
- Part 2: Aldafermin 0.3 mg: Participants who received a single subcutaneous injection of aldafermin 0.3 mg. The first dose (Day 1) and doses at Weeks 1, 2, 4, 8, and 12 were self-administered in the clinic, with all other doses through Week 12 self-administered at home.
- Part 2: Aldafermin 1.0 mg: Participants who received a single subcutaneous injection of aldafermin 1.0 mg. The first dose (Day 1) and doses at Weeks 1, 2, 4, 8, and 12 were self-administered in the clinic, with all other doses through Week 12 self-administered at home.
- Part 2: Aldafermin 3.0 mg: Participants who received a single subcutaneous injection of aldafermin 3.0 mg. The first dose (Day 1) and doses at Weeks 1, 2, 4, 8, and 12 were self-administered in the clinic, with all other doses through Week 12 self-administered at home.
- Part 2: Aldafermin 1.0 mg (Cohort 4): Participants who received a single subcutaneous injection of aldafermin 1.0 mg (Cohort 4). The first dose (Day 1) and doses at Weeks 1, 2, 4, 8, and 12 were self-administered in the clinic, with all other doses through Week 12 self-administered at home.
- Part 3: Aldafermin 1.0 mg: Participants who were randomized to receive a single subcutaneous injection of aldafermin 1.0 mg. The first dose (Day 1) and doses at Weeks 1, 2, 4, 8, and 12 were self-administered in the clinic, with all other doses through Week 12 self-administered at home.
Period: Part 1
Arm/Group | Part 1: Aldafermin 3.0 mg | Part 1: Aldafermin 6.0 mg | Part 1: Placebo | Part 2: Aldafermin 0.3 mg | Part 2: Aldafermin 1.0 mg | Part 2: Aldafermin 3.0 mg | Part 2: Aldafermin 1.0 mg (Cohort 4) | Part 3: Aldafermin 1.0 mg | Part 3: Placebo
Started | 27 | 28 | 27 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 25 | 24 | 23 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 2 | 4 | 4 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 2 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrew informed consent | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Participant moved out of state | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Participant enrolled in another clinical trial | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 2
Arm/Group | Part 1: Aldafermin 3.0 mg | Part 1: Aldafermin 6.0 mg | Part 1: Placebo | Part 2: Aldafermin 0.3 mg | Part 2: Aldafermin 1.0 mg | Part 2: Aldafermin 3.0 mg | Part 2: Aldafermin 1.0 mg (Cohort 4) | Part 3: Aldafermin 1.0 mg | Part 3: Placebo
Started (Patients enrolled in Part 1 did not participate in Part 2.) | 0 (Patients enrolled in Part 1 Aldafermin 3.0 mg did not participate in Part 2.) | 0 (Patients enrolled in Part 1 Aldafermin 6.0 mg did not participate in Part 2.) | 0 (Patients enrolled in Part 1 Placebo did not participate in Part 2.) | 23 (Patients enrolled in Part 1 did not participate in Part 2.) | 21 (Patients enrolled in Part 1 did not participate in Part 2.) | 22 (Patients enrolled in Part 1 did not participate in Part 2.) | 28 (Patients enrolled in Part 1 did not participate in Part 2.) | 0 (Patients enrolled in Part 3 did not participate in Part 2.) | 0 (Patients enrolled in Part 3 did not participate in Part 2.)
Completed | 0 | 0 | 0 | 21 | 20 | 19 | 25 | 0 | 0
Not Completed | 0 | 0 | 0 | 2 | 1 | 3 | 3 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 0
Not completed — Withdrew informed consent | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Not completed — Inability to comply with protocol | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Early end of treatment secondary to cardiac arrest and subsequently lost to follow up | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Period: Part 3
Arm/Group | Part 1: Aldafermin 3.0 mg | Part 1: Aldafermin 6.0 mg | Part 1: Placebo | Part 2: Aldafermin 0.3 mg | Part 2: Aldafermin 1.0 mg | Part 2: Aldafermin 3.0 mg | Part 2: Aldafermin 1.0 mg (Cohort 4) | Part 3: Aldafermin 1.0 mg | Part 3: Placebo
Started (Patients enrolled in Part 2 did not participate in Part 3.) | 0 | 0 | 0 | 0 (Patients enrolled in Part 2 did not participate in Part 3.) | 0 (Patients enrolled in Part 2 did not participate in Part 3.) | 0 (Patients enrolled in Part 2 did not participate in Part 3.) | 0 (Patients enrolled in Part 2 did not participate in Part 3.) | 53 (Patients enrolled in Part 2 did not participate in Part 3.) | 25 (Patients enrolled in Part 2 did not participate in Part 3.)
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 49 | 20
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 5
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Withdrew informed consent | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 2
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2

BASELINE CHARACTERISTICS:
Population: Baseline characteristics were reported from the Safety Population.
Groups:
- Part 3: Aldafermin 1.0 mg: Participants who were randomized to receive a single subcutaneous injection of aldafermin 1.0 mg. The first dose (Day 1) and doses at Weeks 1, 2, 4, 6, 8, 12, 18, and 24 were self-administered in the clinic, with all other doses throughout the treatment period self-administered at home.
- Part 3: Placebo: Participants who were randomized to receive a single subcutaneous injection of placebo. The first dose (Day 1) and doses at Weeks 1, 2, 4, 6, 8, 12, 18, and 24 were self-administered in the clinic, with all other doses throughout the treatment period self-administered at home.
- Total: Total of all reporting groups
Arm/Group | Part 1: Aldafermin 3.0 mg | Part 1: Aldafermin 6.0 mg | Part 1: Placebo | Part 2: Aldafermin 0.3 mg | Part 2: Aldafermin 1.0 mg | Part 2: Aldafermin 3.0 mg | Part 2: Aldafermin 1.0 mg (Cohort 4) | Part 3: Aldafermin 1.0 mg | Part 3: Placebo | Total
Number analyzed (Participants) | 27 | 28 | 27 | 23 | 21 | 22 | 28 | 53 | 25 | 254
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 26 | 26 | 23 | 22 | 17 | 18 | 26 | 45 | 23 | 226
  >=65 years | 1 | 2 | 4 | 1 | 4 | 4 | 2 | 8 | 2 | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.0 (7.1) | 56.4 (7.8) | 52.8 (11.3) | 43.0 (11.7) | 51.5 (11.3) | 51.5 (11.7) | 49.8 (10.0) | 53.2 (12.1) | 54.1 (9.7) | 51.9 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 16 | 20 | 13 | 18 | 18 | 20 | 26 | 16 | 163
  Male | 11 | 12 | 7 | 10 | 3 | 4 | 8 | 27 | 9 | 91
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 3 | 0 | 6
  Black | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 2 | 5
  White | 25 | 24 | 25 | 23 | 21 | 22 | 26 | 46 | 22 | 234
  Pacific Islander | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Other | 1 | 2 | 0 | 0 | 0 | 0 | 1 | 3 | 1 | 8

OUTCOME MEASURES:

1. Primary Outcome: Change in Absolute Liver Fat Content (Part 1)
Description: Absolute liver fat content was assessed using magnetic resonance imaging (MRI).
Time Frame: Up to Week 12
Population: Absolute liver fat content was assessed in participants with available data in the Efficacy Population.
Measure: Least Squares Mean (Standard Error); unit: percent of liver fat
Arm/Group | Part 1: Aldafermin 3.0 mg | Part 1: Aldafermin 6.0 mg | Part 1: Placebo
Number analyzed (Participants) | 27 | 28 | 27
percent of liver fat | -9.68 (0.98) | -11.91 (1.00) | -0.85 (0.99)
Statistical Analysis 1: Comparison: Part 1: Aldafermin 3.0 mg vs Part 1: Placebo; The absolute change in liver fat content from baseline to Week 12 was compared between treatment groups using an ANCOVA model with treatment group and diabetic status as cofactors and baseline endpoint and baseline alanine aminotransferase (ALT) as covariates; Test type: Superiority; p < 0.001, t-test, 2 sided — p-values are adjusted using a stepdown-Bonferroni method to adjust for multiple testing; Difference in least squares means = -8.84, 96% CI 2-sided [-12.09 to -5.59], Standard Error of Mean 1.37
Statistical Analysis 2: Comparison: Part 1: Aldafermin 6.0 mg vs Part 1: Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.001, t-test, 2 sided — p-values are adjusted using a stepdown-Bonferroni method to adjust for multiple testing; Difference in least squares means = -11.06, 96% CI 2-sided [-14.39 to -7.74], Standard Error of Mean 1.40
Statistical Analysis 3: Comparison: Part 1: Aldafermin 3.0 mg vs Part 1: Aldafermin 6.0 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.112, t-test, 2 sided; Difference in least squares means = -2.22, 96% CI 2-sided [-5.11 to 0.67], Standard Error of Mean 1.38

2. Primary Outcome: Change in Absolute Liver Fat Content (Part 2)
Description: Absolute liver fat content was assessed using magnetic resonance imaging proton density fat fraction (MRI-PDFF).
Time Frame: Up to Week 12
Population: Absolute liver fat content was assessed in participants with available data in the Efficacy Population.
Measure: Least Squares Mean (Standard Error); unit: percent of liver fat
Arm/Group | Part 2: Aldafermin 0.3 mg | Part 2: Aldafermin 1.0 mg | Part 2: Aldafermin 3.0 mg | Part 2: Aldafermin 1.0 mg (Cohort 4)
Number analyzed (Participants) | 23 | 21 | 20 | 25
percent of liver fat | -4.95 (1.07) | -10.69 (1.09) | -11.55 (1.08) | -10.85 (1.01)
Statistical Analysis 1: Comparison: Part 2: Aldafermin 0.3 mg vs Part 2: Aldafermin 1.0 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.0001, t-test, 2 sided; Difference in least squares means = -5.73, 95% CI 2-sided [-8.48 to -2.99], Standard Error of Mean 1.38
Statistical Analysis 2: Comparison: Part 2: Aldafermin 0.3 mg vs Part 2: Aldafermin 3.0 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.0001, t-test, 2 sided; Difference in least squares means = -6.60, 95% CI 2-sided [-9.41 to -3.79], Standard Error of Mean 1.41
Statistical Analysis 3: Comparison: Part 2: Aldafermin 1.0 mg vs Part 2: Aldafermin 3.0 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.5467, t-test, 2 sided; Difference in least squares means = -0.87, 95% CI 2-sided [-3.71 to 1.98], Standard Error of Mean 1.43
Statistical Analysis 4: Comparison: Part 2: Aldafermin 0.3 mg vs Part 2: Aldafermin 1.0 mg (Cohort 4); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.0001, t-test, 2 sided; Difference in least squares means = -5.90, 95% CI 2-sided [-8.55 to -3.25], Standard Error of Mean 1.33
Statistical Analysis 5: Comparison: Part 2: Aldafermin 1.0 mg vs Part 2: Aldafermin 1.0 mg (Cohort 4); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.9037, t-test, 2 sided; Difference in least squares means = -0.17, 95% CI 2-sided [-2.89 to 2.55], Standard Error of Mean 1.37
Statistical Analysis 6: Comparison: Part 2: Aldafermin 3.0 mg vs Part 2: Aldafermin 1.0 mg (Cohort 4); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.6134, t-test, 2 sided; Difference in least squares means = 0.70, 95% CI 2-sided [-2.05 to 3.45], Standard Error of Mean 1.38

3. Primary Outcome: Change in Absolute Liver Fat Content (Part 3)
Description: Absolute liver fat content was measured by magnetic resonance imaging proton density fat fraction (MRI-PDFF).
Time Frame: Up to Week 24
Population: Absolute liver fat content was assessed in participants with available data in the Efficacy Population.
Measure: Least Squares Mean (Standard Error); unit: percent of liver fat
Arm/Group | Part 3: Aldafermin 1.0 mg | Part 3: Placebo
Number analyzed (Participants) | 51 | 22
percent of liver fat | -7.70 (0.82) | -2.73 (1.29)
Statistical Analysis 1: Comparison: Part 3: Aldafermin 1.0 mg vs Part 3: Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.0018, t-test, 2 sided; Difference in least squares means = -4.97, 95% CI 2-sided [-8.03 to -1.91], Standard Error of Mean 1.53

4. Secondary Outcome: Percentage Change in Liver Fat Content (Part 1)
Description: Percentage change in liver fat content was assessed using magnetic resonance imaging (MRI).
Time Frame: Up to Week 12
Population: Percentage change in liver fat content was assessed in the Efficacy Population.
Measure: Least Squares Mean (Standard Error); unit: percentage change of liver fat content
Arm/Group | Part 1: Aldafermin 3.0 mg | Part 1: Aldafermin 6.0 mg | Part 1: Placebo
Number analyzed (Participants) | 27 | 28 | 27
percentage change of liver fat content | -47.98 (5.79) | -60.09 (5.92) | -2.57 (5.85)

5. Secondary Outcome: Change in Absolute Liver Fat Content (Part 2)
Description: Absolute liver fat content was assessed using magnetic resonance imaging proton density fat fraction (MRI-PDFF).
Time Frame: Up to Week 18
Population: Absolute liver fat content was assessed in participants with available data in the Efficacy Population.
Measure: Least Squares Mean (Standard Error); unit: percent of liver fat
Arm/Group | Part 2: Aldafermin 0.3 mg | Part 2: Aldafermin 1.0 mg | Part 2: Aldafermin 3.0 mg | Part 2: Aldafermin 1.0 mg (Cohort 4)
Number analyzed (Participants) | 23 | 21 | 20 | 26
percent of liver fat
  Week 6 | -4.15 (0.93) | -8.21 (0.97) | -10.38 (0.94) | -8.36 (0.87)
  Week 18: number analyzed (Participants) | 20 | 21 | 19 | 24
  Week 18 | -4.51 (1.17) | -3.87 (1.14) | -7.67 (1.15) | -5.72 (1.07)

6. Secondary Outcome: Percentage Change in Liver Fat Content (Part 2)
Description: Percentage change in liver fat content was assessed using magnetic resonance imaging proton density fat fraction (MRI-PDFF).
Time Frame: Up to Week 18
Population: Percentage change in liver fat content was assessed in participants with available data in the Efficacy Population.
Measure: Least Squares Mean (Standard Error); unit: percentage change of liver fat content
Arm/Group | Part 2: Aldafermin 0.3 mg | Part 2: Aldafermin 1.0 mg | Part 2: Aldafermin 3.0 mg | Part 2: Aldafermin 1.0 mg (Cohort 4)
Number analyzed (Participants) | 23 | 21 | 22 | 28
percentage change of liver fat content
  Week 6: number analyzed (Participants) | 23 | 20 | 22 | 28
  Week 6 | -24.95 (4.94) | -42.90 (5.19) | -58.72 (5.01) | -45.92 (4.63)
  Week 12: number analyzed (Participants) | 23 | 21 | 22 | 25
  Week 12 | -29.09 (5.32) | -55.10 (5.42) | -63.84 (5.41) | -57.85 (5.04)
  Week 18: number analyzed (Participants) | 20 | 21 | 19 | 24
  Week 18 | -22.58 (6.66) | -17.70 (6.44) | -40.79 (6.55) | -29.03 (6.07)

7. Secondary Outcome: Change in Absolute Liver Fat Content (Part 3)
Description: Absolute liver fat content was measured by magnetic resonance imaging proton density fat fraction (MRI-PDFF).
Time Frame: Up to Week 30
Population: Absolute liver fat content was assessed in the Efficacy Population in participants with available data.
Measure: Least Squares Mean (Standard Error); unit: percent of liver fat
Arm/Group | Part 3: Aldafermin 1.0 mg | Part 3: Placebo
Number analyzed (Participants) | 52 | 24
percent of liver fat
  Week 6 | -6.54 (0.59) | -0.93 (0.89)
  Week 12: number analyzed (Participants) | 51 | 22
  Week 12 | -8.43 (0.74) | -1.89 (1.14)
  Week 30: number analyzed (Participants) | 49 | 21
  Week 30 | -3.04 (0.77) | -2.05 (1.19)

8. Secondary Outcome: Percentage Change in Liver Fat Content (Part 3)
Description: as for outcome 6
Time Frame: Up to Week 30
Population: Percentage change in liver fat content was assessed in participants with available data in the Efficacy Population.
Measure: Least Squares Mean (Standard Error); unit: percentage change of liver fat content
Arm/Group | Part 3: Aldafermin 1.0 mg | Part 3: Placebo
Number analyzed (Participants) | 52 | 24
percentage change of liver fat content
  Week 6 | -36.59 (3.22) | -2.17 (4.81)
  Week 12: number analyzed (Participants) | 51 | 22
  Week 12 | -45.27 (4.26) | -6.88 (6.60)
  Week 24: number analyzed (Participants) | 50 | 21
  Week 24 | -38.76 (5.03) | -13.10 (7.89)
  Week 30: number analyzed (Participants) | 49 | 21
  Week 30 | -11.22 (4.91) | -9.99 (7.59)

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events were collected from Screening (Day -28 to Day -1) up to Week 30.
Arm/Group | Part 1: Aldafermin 3.0 mg | Part 1: Aldafermin 6.0 mg | Part 1: Placebo | Part 2: Aldafermin 0.3 mg | Part 2: Aldafermin 1.0 mg | Part 2: Aldafermin 3.0 mg | Part 2: Aldafermin 1.0 mg (Cohort 4) | Part 3: Aldafermin 1.0 mg | Part 3: Placebo
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/28 | 0/27 | 0/23 | 0/21 | 0/22 | 0/28 | 0/53 | 0/25
Serious Adverse Events (participants affected / at risk) | 1/27 | 0/28 | 0/27 | 0/23 | 1/21 | 4/22 | 1/28 | 2/53 | 3/25
Other Adverse Events (participants affected / at risk) | 26/27 | 27/28 | 23/27 | 20/23 | 19/21 | 21/22 | 27/28 | 46/53 | 22/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: Aldafermin 3.0 mg (N=27) | Part 1: Aldafermin 6.0 mg (N=28) | Part 1: Placebo (N=27) | Part 2: Aldafermin 0.3 mg (N=23) | Part 2: Aldafermin 1.0 mg (N=21) | Part 2: Aldafermin 3.0 mg (N=22) | Part 2: Aldafermin 1.0 mg (Cohort 4) (N=28) | Part 3: Aldafermin 1.0 mg (N=53) | Part 3: Placebo (N=25)
Acute pancreatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac arrest (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vertigo positional (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Renal mass (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Accelerated hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Mental status changes (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Suicidal ideation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Post procedural complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: Aldafermin 3.0 mg (N=27) | Part 1: Aldafermin 6.0 mg (N=28) | Part 1: Placebo (N=27) | Part 2: Aldafermin 0.3 mg (N=23) | Part 2: Aldafermin 1.0 mg (N=21) | Part 2: Aldafermin 3.0 mg (N=22) | Part 2: Aldafermin 1.0 mg (Cohort 4) (N=28) | Part 3: Aldafermin 1.0 mg (N=53) | Part 3: Placebo (N=25)
Loose stools (Gastrointestinal disorders) | 7 | 5 | 2 | 1 | 3 | 5 | 6 | 0 | 0
Nausea (Gastrointestinal disorders) | 8 | 3 | 1 | 2 | 6 | 6 | 12 | 5 | 6
Diarrhea (Gastrointestinal disorders) | 2 | 3 | 4 | 0 | 3 | 2 | 8 | 15 | 6
Vomiting (Gastrointestinal disorders) | 2 | 5 | 0 | 2 | 3 | 2 | 6 | 3 | 1
Abdominal pain (Gastrointestinal disorders) | 3 | 3 | 0 | 1 | 1 | 1 | 2 | 2 | 1
Bloating (Gastrointestinal disorders) | 1 | 4 | 0 | 0 | 2 | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 3 | 1 | 1 | 1 | 1 | 1 | 5 | 3 | 1
Nausea aggravated (Gastrointestinal disorders) | 2 | 2 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Abdominal bloating (Gastrointestinal disorders) | 2 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Diarrhea aggravated (Gastrointestinal disorders) | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hemorrhoids (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
RUQ pain (Gastrointestinal disorders) | 2 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Soft stools (Gastrointestinal disorders) | 1 | 2 | 0 | 1 | 1 | 0 | 0 | 0 | 0
GERD (Gastrointestinal disorders) | 2 | 0 | 0 | 1 | 1 | 0 | 0 | 4 | 0
Increased frequency of defecation (Gastrointestinal disorders) | 2 | 0 | 0 | 1 | 2 | 1 | 0 | 0 | 0
Stomach cramps (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Injection site erythema (General disorders) | 6 | 11 | 2 | 0 | 2 | 0 | 1 | 0 | 0
Injection site reaction (General disorders) | 3 | 4 | 0 | 1 | 0 | 1 | 1 | 2 | 0
Injection site bruising (General disorders) | 2 | 0 | 3 | 1 | 0 | 0 | 0 | 3 | 0
Injection site pruritus (General disorders) | 2 | 3 | 0 | 0 | 1 | 0 | 3 | 1 | 0
Fatigue (General disorders) | 0 | 2 | 2 | 3 | 3 | 1 | 6 | 3 | 4
Injection site pain (General disorders) | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Injection site swelling (General disorders) | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 3 | 5 | 5 | 5 | 4 | 4 | 4 | 7 | 9
Dysgeusia (Nervous system disorders) | 1 | 1 | 2 | 0 | 1 | 0 | 0 | 1 | 2
Dizziness (Nervous system disorders) | 2 | 1 | 0 | 0 | 1 | 0 | 4 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 2 | 2 | 2 | 1 | 0 | 1 | 1 | 1
Sinusitis (Infections and infestations) | 2 | 1 | 1 | 1 | 1 | 0 | 2 | 4 | 2
Urinary tract infection (Infections and infestations) | 2 | 2 | 0 | 0 | 1 | 4 | 3 | 2 | 2
Nasopharyngitis (Infections and infestations) | 0 | 0 | 2 | 0 | 1 | 0 | 5 | 2 | 1
Increased appetite (Metabolism and nutrition disorders) | 2 | 4 | 0 | 0 | 2 | 1 | 1 | 1 | 0
Weight decreased (Investigations) | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1
Weight increased (Investigations) | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 0 | 1 | 0 | 0 | 0 | 2 | 2 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2 | 1 | 0 | 1 | 0 | 4 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0 | 2 | 1 | 1 | 2 | 1
Hypertension (Vascular disorders) | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 2 | 2
Haematuria (Renal and urinary disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal cramp (Gastrointestinal disorders) | 1 | 1 | 0 | 1 | 0 | 0 | 2 | 0 | 0
Emesis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Frequent bowel movements (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 3 | 0
Stool discoloration (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Low density lipoprotein increased (Investigations) | 1 | 0 | 0 | 9 | 15 | 9 | 13 | 0 | 0
Blood cholesterol increased (Investigations) | 0 | 0 | 0 | 0 | 2 | 4 | 7 | 0 | 0
Glycosylated hemoglobin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 1 | 2 | 1 | 1 | 2 | 0
Influenza (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 4 | 4 | 6 | 1 | 0
Chest pain (General disorders) | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 4 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 0 | 2 | 4 | 2 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 4 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 2 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 2 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 1 | 1 | 2 | 0 | 0 | 3 | 0
Seasonal allergy (Immune system disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 2 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 3
Oedema peripheral (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 3
Influenza like illness (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 2
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 5
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 1 | 1 | 0 | 1 | 2
Diarrhoea (Gastrointestinal disorders) | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 15 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-03-29): https://cdn.clinicaltrials.gov/large-docs/16/NCT02443116/Prot_000.pdf
  • Statistical Analysis Plan (2019-10-01): https://cdn.clinicaltrials.gov/large-docs/16/NCT02443116/SAP_001.pdf